CLINICAL TRIAL: NCT01047852
Title: Sequential and Early Used of Noninvasive Ventilation After Extubation in Hypercapnic Patients or in Patients With Chronic Respiratory Disorders
Brief Title: Noninvasive Ventilation After Extubation in Hypercapnic Patients
Acronym: VHYPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2009/10
Record Dates: First submitted 2010-01-05; First posted 2010-01-13 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Respiratory Failure
Keywords: chronic respiratory disorders; hypercapnic respiratory failure; noninvasive ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIV (Experimental)
  Interventions: Procedure: Noninvasive ventilation
- Control (No Intervention)

INTERVENTIONS:
Procedure: Noninvasive ventilation — NIV will be delivered using a sequential mode (a minimum of 1 hour every 3 hours) immediately after extubation for a schedule period of 48 h after extubation. In between NIV courses ((NIV-free periods) O2 will be administered through nasal cannula in order to obtain a SaO2 ≥ 90%. Afterward, NIV will be withdraw and oxygen will be administered by nasal cannula
  Arms: NIV

SUMMARY:
The purpose of this study is to assess the efficacy of noninvasive ventilation (NIV) in the prevention of extubation failure and mortality in patients with either chronic respiratory disorders or hypercapnic respiratory failure during spontaneous breathing.

DETAILED DESCRIPTION:
Reintubation, which occurs in 6 to 23% within 48 to 72 hours after planned extubation, is a relevant consequence of respiratory failure after extubation. Patients with chronic respiratory disorders and invasively mechanically ventilated in intensive care unit, often exhibit hypercapnia, during breathing trial prior extubation. This is associated to increased incidence of extubation failure and mortality. Although the need for reintubation may be a marker of increased severity of illness, this is an independent risk factor for nosocomial pneumonia, increased hospital stay and mortality. NIV does not seem to be beneficial in avoiding reintubation when these patients have developed respiratory failure. However, a recent randomised study demonstrated that the early use of NIV averted respiratory failure after extubation in patients at increased risk. The patients were considered at risk if they had at least one of the following criteria: age > 65 years, cardiac failure, increased severity assessed by an Acute Physiologic and Chronic Health Evaluation score > 12. But, the beneficial effects of NIV on survival appear to be restricted to patients with chronic respiratory disorders and hypercapnia during the spontaneous breathing trial. So the beneficial effects of NIV should be confirmed in a trial in this specific population. We planned to conduct a study evaluating the efficacy of NIV in the prevention of extubation failure and mortality in these patients. If no signs of respiratory failure appeared after 120 min of a spontaneous breathing trial, patients will be extubated and randomly allocated after extubation to NIV group or control group. The clinical follow-up will be as follow: the incidence of extubation failure, the reintubation, the ICU and hospital mortality, 28-day survival, the complications associated to mechanical ventilation, ICU and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients intubated for 48 hours or more
* Patients with Chronic respiratory disorders
* And/or hypercapnic respiratory failure during successful spontaneous breathing trial

Exclusion Criteria:

* Face or cranial trauma or surgery
* Home noninvasive ventilation
* Recent gastric or oesophageal surgery
* Tracheostomy or other upper airway disorders
* Upper gastrointestinal bleeding
* Excess respiratory secretions
* Lack of collaboration
* Do not resuscitate order or any decision to limit therapeutic effort in the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory failure after extubation | 2 days

SECONDARY OUTCOMES:
Incidence of reintubation | 2 months
Length of stay in Intensive Care Unit | 2 months
Hospital mortality | 2 months
Survival | 28th day
Survival | 90th day
Incidence of complications associated to mechanical ventilation | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VARGAS, MD, Principal Investigator — University Hospital, Bordeaux, France; Olivier GUISSET, MD, Principal Investigator — University Hospital, Bordeaux, France; Marc CLAVEL, MD, Principal Investigator — University Hospital, Limoges, France; Pascale SANCHEZ, MD, Principal Investigator — University Hospital, Toulouse, France; Sylvain GARNIER, MD, Principal Investigator — Hospital, Libourne, France; Aissa KHERCHACHE, MD, Principal Investigator — Hospital, Agen, France; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux, France
Locations (6):
- France (6):
  - Hospital, Agen
  - Saint-André Hospital, Bordeaux
  - Pellegrin Hospital, Recovery Unit, Bordeaux
  - Hospital, Libourne
  - University Hospital, Limoges
  - University Hospital, Toulouse

REFERENCES:
- [Derived] Vargas F, Clavel M, Sanchez-Verlan P, Garnier S, Boyer A, Bui HN, Clouzeau B, Sazio C, Kerchache A, Guisset O, Benard A, Asselineau J, Gauche B, Gruson D, Silva S, Vignon P, Hilbert G. Intermittent noninvasive ventilation after extubation in patients with chronic respiratory disorders: a multicenter randomized controlled trial (VHYPER). Intensive Care Med. 2017 Nov;43(11):1626-1636. doi: 10.1007/s00134-017-4785-1. Epub 2017 Apr 9. PMID 28393258